CLINICAL TRIAL: NCT06410027
Title: Effects of Pain Neuroscience Education and Virtual Reality in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Torres Sánchez, PT, PhD, Principal investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DLCRV-01
Record Dates: First submitted 2024-04-19; First posted 2024-05-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2024-04

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education + Virtual Reality + Therapeutic Exercise (Experimental): 1-hour pain neuroscience education session + 30-minutes exposure to exercise with virtual reality + Therapeutic Exercise
  Interventions: Other: Pain Neuroscience Education + Virtual Reality + Therapeutic Exercise
- Therapeutic Exercise (Active Comparator): Therapeutic Exercise
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Other: Pain Neuroscience Education + Virtual Reality + Therapeutic Exercise — Patients will receive 1-hour pain neuroscience education session + 30-minutes exposure to exercise with virtual reality + therapeutic exercise
  Arms: Pain Neuroscience Education + Virtual Reality + Therapeutic Exercise
Other: Therapeutic Exercise — Patients will receive therapeutic exercise
  Arms: Therapeutic Exercise

SUMMARY:
The objective of our study is to evaluate the effects of a therapeutic intervention including

1-hour of pain neuroscience education session, 30-minutes of exposure to exercise with virtual realit and therapeutic exercise in patients with chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain is the world's leading cause of years of life lived with disability. Negative thoughts and beliefs about pain experienced can lead to pain avoidance behaviours. Fear of movement is a common behaviour in this type of patients and is associated with avoidance of exercise. Virtual reality is a powerful distraction technique as it directs the patient's attention to an external stimulus rather than pain or body movement. Therefore, it can be beneficial to avoid some pain-related problems, such as kinesiophobia and inactivity. Moreover, pain neuroscience education aim to reconceptualise pain perceptions, beliefs, and avoidance behaviours. Then, the use of these interventions may be beneficial in the treatment of patients with chronic low back pain.

The objective of this study is to evaluate the effects of a therapeutic intervention using pain neuroscience education and virtual reality in patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain (≥ 3 months)
* Adults (≥ 18 years and less than 65 years)
* Score ≤18 points in Pain Detect Scale
* Wish to participate in the study and sign the informed consent
* Speaking Spanish

Exclusion Criteria:

* Neuropathic pain (score >18 in Pain Detect Scale)
* Physical or psychological pathology of any kind that imply an inability to understand the necessary instructions to carry out the study will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Pre-intervention
  To assess pain intensity using the Numeric Pain Rating Scale. Scores range from 0 (no pain) to 10 (worst pain imaginable). Higher scores indicate greater intensity.
Pain Intensity | 48-72h after the intervention
  To assess pain intensity using the Numeric Pain Rating Scale. Scores range from 0 (no pain) to 10 (worst pain imaginable). Higher scores indicate greater intensity.
Pain Intensity and Interference | Pre-intervention
  To assess pain intensity and interference using the Brief Pain Inventory (BPI). Scores range from 0 (no pain/does not interfere) to 10 (worst pain imaginable/completely interferes). Higher scores indicate greater intensity and interference.
Pain Intensity and Interference | 48-72h after the intervention
  To assess pain intensity and interference using the Brief Pain Inventory (BPI). Scores range from 0 (no pain/does not interfere) to 10 (worst pain imaginable/completely interferes). Higher scores indicate greater intensity and interference.
Neurophysiology of Pain | Pre-intervention
  To assess neurophysiology of pain using the Neurophysiology of Pain Questionnaire (NPQ). Scores range from 0 to 13 (sum of all correct items).
Neurophysiology of Pain | 48-72h after the intervention
  To assess neurophysiology of pain using the Neurophysiology of Pain Questionnaire (NPQ). Scores range from 0 to 13 (sum of all correct items).
Pain-Self Efficacy | Pre-intervention
  To assess pain-self efficacy using 10 items Pain Self-Efficacy Questionnaire (10-PSEQ). Scores range from 0 (not at all confident) and 6 (completely confident). A total score is calculated by summing the scores for each of the 10 items, yielding a maximum possible score of 60. Higher scores reflect stronger self-efficacy beliefs.
Pain-Self Efficacy | 48-72h after the intervention
  To assess pain-self efficacy using 10 items Pain Self-Efficacy Questionnaire (10-PSEQ). Scores range from 0 (not at all confident) and 6 (completely confident). A total score is calculated by summing the scores for each of the 10 items, yielding a maximum possible score of 60. Higher scores reflect stronger self-efficacy beliefs.
Awareness, Consciousness, Vigilance and Observation of pain | Pre-intervention
  To assess awareness, consciousness, vigilance and observation of pain using the Pain Vigilance and Awareness Questionnaire (PVAQ). Scores range from 0 (never) to 5 (always). The total questionnaire scores range between 0 and 80. Higher scores indicate greater awareness, consciousness, vigilance and observation of pain.
Awareness, Consciousness, Vigilance and Observation of pain | 48-72h after the intervention
  To assess awareness, consciousness, vigilance and observation of pain using the Pain Vigilance and Awareness Questionnaire (PVAQ). Scores range from 0 (never) to 5 (always). The total questionnaire scores range between 0 and 80. Higher scores indicate greater awareness, consciousness, vigilance and observation of pain.
Catastrophizing of pain | Pre-intervention
  To assess catastrophizing of pain using the Pain Catastrophizing Scale (PCS). Scores range from 0 (nothing at all) to 4 (all the time). The final score range between 0 and 52 points, with higher scores indicating greater levels of catastrophism.
Catastrophizing of pain | 48-72h after the intervention
  To assess catastrophizing of pain using the Pain Catastrophizing Scale (PCS). Scores range from 0 (nothing at all) to 4 (all the time). The final score range between 0 and 52 points, with higher scores indicating greater levels of catastrophism.
Fear and avoidance beliefs | Pre-intervention
  To assess fear and avoidance beliefs using Fear and Avoidance Beliefs Questionnaire (FABQ). Scores range from 0 (totally disagree) to 6 (totally agree). The total score range from 0 to 96, with a higher value reflecting a higher degree of fear avoidance beliefs.
Fear and avoidance beliefs | 48-72h after the intervention
  To assess fear and avoidance beliefs using Fear and Avoidance Beliefs Questionnaire (FABQ). Scores range from 0 (totally disagree) to 6 (totally agree). The total score range from 0 to 96, with a higher value reflecting a higher degree of fear avoidance beliefs.
Kinesiophobia | Pre-intervention
  To assess kinesiophobia using the TAMPA Scale of Kinesiophobia (TSK). Scores range from 1 (totally disagree) to 4 (totally agree). The final score can range between 11 and 44 points, with higher scores indicating greater perceived kinesiophobia.
Kinesiophobia | 48-72h after the intervention
  To assess kinesiophobia using the TAMPA Scale of Kinesiophobia (TSK). Scores range from 1 (totally disagree) to 4 (totally agree). The final score can range between 11 and 44 points, with higher scores indicating greater perceived kinesiophobia.
Health-related Quality of Life | Pre-intervention
  To assess health-related quality of life using the EuroQol-5D. Total score range from 1 (best health status) to 0 (death). The second part of the euroqol-5d is visual analogue scale that goes from 0 (worst state of health imaginable) to 100 (best state of health imaginable).
Health-related Quality of Life | 48-72h after the intervention
  To assess health-related quality of life using the EuroQol-5D. Total score range from 1 (best health status) to 0 (death). The second part of the euroqol-5d is visual analogue scale that goes from 0 (worst state of health imaginable) to 100 (best state of health imaginable).
Algometry | Pre-intervention
  To assess pain pressure threshold using algometer Force One FPIX 50. With the patient sitting in a comfortable position, the different bilateral points where sensitivity is to be evaluated will be marked on the skin. The chosen points are the nail phalanx of the thumb, the gracilis muscle at its insertion, the second rib, the supraspinatus muscle, and the middle portion of the trapezius. In the order described, pressure will be applied perpendicular to the point at a speed of 1 kg/sec until the patient stops the test when the sensation is no longer just "contact", but "discomfort". 3 repetitions will be done, leaving 1 minute between each of them and the average value will be calculated.
Algometry | 48-72h after the intervention
  To assess pain pressure threshold using algometer Force One FPIX 50. With the patient sitting in a comfortable position, the different bilateral points where sensitivity is to be evaluated will be marked on the skin. The chosen points are the nail phalanx of the thumb, the gracilis muscle at its insertion, the second rib, the supraspinatus muscle, and the middle portion of the trapezius. In the order described, pressure will be applied perpendicular to the point at a speed of 1 kg/sec until the patient stops the test when the sensation is no longer just "contact", but "discomfort". 3 repetitions will be done, leaving 1 minute between each of them and the average value will be calculated.
Temporal summation | Pre-intervention
  To assess temporal summation using algometer Force One FPIX 50. The pressure pain threshold will be evaluated in the flexor digitorum muscle in both forearms. The average of both measurements will be calculated. A series of 15 stimuli will be presented to one arm at an interstimulus interval of 3s and then to the other arm at an interstimulus interval of 5s, separated by a 30s interseries interval. After a short break, the series of stimuli will be repeated in reverse order. Patients will be instructed to provide numerical ratings of the magnitude of the sensation experienced during the first, fifth, tenth, and fifteenth period after repeated brief taps. They will be also asked to report on the magnitude of after-sensations present 15 and 60 s after the last stimulus in each series.
Temporal summation | 48-72h after the intervention
  To assess temporal summation using algometer Force One FPIX 50. The pressure pain threshold will be evaluated in the flexor digitorum muscle in both forearms. The average of both measurements will be calculated. A series of 15 stimuli will be presented to one arm at an interstimulus interval of 3s and then to the other arm at an interstimulus interval of 5s, separated by a 30s interseries interval. After a short break, the series of stimuli will be repeated in reverse order. Patients will be instructed to provide numerical ratings of the magnitude of the sensation experienced during the first, fifth, tenth, and fifteenth period after repeated brief taps. They will be also asked to report on the magnitude of after-sensations present 15 and 60 s after the last stimulus in each series.
Chronic pain modulation | Pre-intervention
  To assess pain modulation using algometer Force One FPIX 50. The pressure pain threshold will be evaluated in the tibialis anterior muscle and the deltoid muscle. Then the conditioning stimulus will be introduced. A clamp will be placed on the earlobe for 60 seconds. When pain VAS of the earlobe become more than 60 mm, pain pressure threshold will be evaluated again.
Chronic pain modulation | 48-72h after the intervention
  To assess pain modulation using algometer Force One FPIX 50. The pressure pain threshold will be evaluated in the tibialis anterior muscle and the deltoid muscle. Then the conditioning stimulus will be introduced. A clamp will be placed on the earlobe for 60 seconds. When pain VAS of the earlobe become more than 60 mm, pain pressure threshold will be evaluated again.
Electromyography | Pre-intervention
  To assess muscular activity using electromyography with Biosignalplux device (Research Kit Biosignalplux, PLUX Wireless Biosignal S.A). A functional task and flexion-relaxion fenomenon will be evaluated.
Electromyography | 48-72h after the intervention
  To assess muscular activity using electromyography with Biosignalplux device (Research Kit Biosignalplux, PLUX Wireless Biosignal S.A). A functional task and flexion-relaxion fenomenon will be evaluated.

SECONDARY OUTCOMES:
Central Sensitization | Pre-intervention
  To identify when a patient's symptoms may be related to central sensitization using Central Sensitization Inventory (CSI). Responses are recorded for the frequency of each symptom on a Likert scale from 0 (never) to 4 (always), resulting in a total possible score of 100. Higher scores are associated with a higher degree of self-reported symptomatology.
Disability | Pre-intervention
  To assess disability using the Oswestry Disability Index (ODI). Total scores range from 0% (no limitation) to 100% (maximum functional limitation).
Physical activity | Pre-intervention
  To assess physical activity using the International Physical Activity Questionnaire. This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in Metabolic Equivalent (MET)-min/week and time spent sitting.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Torres Sánchez, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Spain